CLINICAL TRIAL: NCT06645743
Title: Clinical and Imaging Features Were Used to Predict the Occurrence of Spread Through Air Space in Stage IA Lung Adenocarcinoma
Brief Title: Retrospective Analysis of Clinical and CT Features to Predict Spread Through Air Space in Stage IA Lung Adenocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: The Third Affiliated Hospital of Kunming Medical College. (Other)
Responsible Party: Principal Investigator, Yantao Yang, doctor, The Third Affiliated Hospital of Kunming Medical College.
Other Study IDs: KYLX2023-137
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Tomography, X-Ray Computed; Spread Through Air Space; Clinical Features; Stage IA Adenocarcinoma of Lung
Keywords: clinical feature; Radiologic characteristic; Lung adenocarcinoma; spread through air space
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spread through air space positive group: The patients in this group were stage IA lung adenocarcinoma patients who met the inclusion and exclusion criteria, and the postoperative pathological results indicated the presence of spread through air space
- spread through air space negative group: The patients in this group were stage IA lung adenocarcinoma patients who met the inclusion and exclusion criteria, and the postoperative pathological results showed no spread through air space

SUMMARY:
The purpose of this study is to provide a basis for the selection of surgical methods for patients with stage IA lung adenocarcinoma. Air cavity dissemination is a poor prognostic factor for patients with stage IA lung adenocarcinoma. We retrospectively collected clinical and imaging data of stage IA lung adenocarcinoma patients. Independent risk factors associated with spread through air space in stage IA lung adenocarcinoma patients were analyzed, so as to predict the occurrence of spread through air space and provide basis for the selection of surgical methods

DETAILED DESCRIPTION:
Referring from Global Cancer Report 2020, lung cancer remains the leading cause of tumor death, with adenocarcinoma as the primary histological subtype. In 2021, the World Health Organization (WHO) proposed a new classification standard for lung cancer, dividing adenocarcinomas into in-situ adenocarcinomas, microinvasive adenocarcinomas, and invasive adenocarcinomas based on their invasive development.

Due to the widespread popularization of early screening for lung cancer, a growing number of IA lung adenocarcinomas cases manifesting as lung nodules have been detected, and surgical resection remains the most critical treatment options for such individuals. With the emergence of relevant research results, sublobectomy has become a preferred method for early stage IA lung adenocarcinoma. However, some individuals with lung adenocarcinoma in stage IA undergoing sublobectomy still have recurrence and metastasis, in which spread through air spaces (STAS) plays vital role.

STAS was formally proposed by WHO in 2015 as a new invasion mode of invasive lung adenocarcinoma. STAS is characterized by pathological micropapillary clusters, solid nests, or isolated cells located beyond the tumor margin, counting one or more, infiltrating the air spaces within the surrounding lung parenchyma and detached from the primary tumor, rather than forming distinct tumor islands. A number of studies have pointed out that STAS is associated with poor prognosis of patients, many researchers continue to favor lobectomy when treating patients with stage IA lung adenocarcinoma exhibiting positive STAS.

Due to the limitations of intraoperative frozen section in predicting STAS, preoperative application of clinical and imaging features in predicting STAS shows great advantages. Former research has suggested that clinical and imaging characteristics can predict occurrence of STAS, despite the difference of results from different studies. Onozato et al. believe that smokers are more likely to develop STAS, which is consistent with the study by Shiono et al. However, Uruga et albelieved that the occurrence of STAS was unrelated to smoking. Warth et al. believed that male lung adenocarcinoma patients were more prone to STAS, while Kadota stated the occurrence of STAS was unrelated to patient gender.

However, the sample size included in these previous studies is small, and the parameters included by various scholars are different, and there is still a lack of large sample studies systematically analyzing clinical and imaging characteristics to predict the spread through air space of stage IA lung adenocarcinoma. Therefore, we plan to carry out this study. Based on a large sample size, the clinical and imaging characteristics of patients with stage IA lung adenocarcinoma were comprehensively analyzed to predict the spread through air space, so as to provide a reference for the selection of surgical methods

ELIGIBILITY:
Inclusion Criteria:

Preoperative CT images reported that the maximum diameter of pulmonary nodules was less than 3 cm

All subjects provided CT imaging obtained from Yunnan Cancer Hospital within a 2-week period prior to surgery

Postoperative pathological diagnosis of invasive lung adenocarcinoma

Remote metastasis was excluded by preoperative imaging (CT, PET-CT, ultrasound, etc.)

Age ≥ 18 years

Exclusion Criteria:

Incomplete collection of medical records, imaging data, or hematology data

Preoperative complications of other malignant tumors

Unclear correspondence between postoperative pathological report and preoperative CT nodule location

Images do not meet analysis conditions due to pulmonary infection or large respiratory motion artifacts

Postoperative pathology revealed two or more nodules classified as infiltrating adenocarcinoma

Prior lung surgery or preoperative neoadjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients diagnosed with Stage IA lung adenocarcinoma after surgery who have undergone preoperative evaluation of clinical and CT imaging at the Third Affiliated Hospital of Kunming Medical University within the past five years
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Predicting Spread Through Air Spaces (STAS) in Stage IA Lung Adenocarcinoma Using Clinical and Imaging Features | Preoperative clinical and imaging data collected within 2 weeks prior to surgery, retrospectively analyzed from patients who underwent surgery within the past 3 years
  This outcome measure assesses the accuracy of using preoperative clinical and CT imaging features to predict the presence of spread through air spaces (STAS) in patients with stage IA lung adenocarcinoma.Measure: Area Under the ROC Curve (AUC), sensitivity, and specificity for the prediction model.

SECONDARY OUTCOMES:
Prognostic Impact of STAS on Recurrence-Free Survival | From the date of surgery to the time of disease recurrence or last follow-up, up to 5 years.
  This outcome measure investigates whether the presence of STAS in stage IA lung adenocarcinoma is associated with recurrence-free survival (RFS).

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — The Third Affiliated Hospital of Kunming Medical University
Locations (1):
- The Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due sharing data is not included in our research institution review board but are available from the corresponding author on reasonable request

REFERENCES:
- See also: Provides global information and statistics on lung cancer — https://www.who.int
- See also: A free search engine providing access to a vast collection of biomedical and life sciences literature, including MEDLINE-indexed articles, covering topics such as medicine, pharmacology, and healthcare research. — https://pubmed.ncbi.nlm.nih.gov
- See also: The Third Affiliated Hospital of Kunming Medical University provides comprehensive cancer care, including surgery, radiotherapy, chemotherapy, and immunotherapy, along with advanced diagnostic and imaging services. — https://www.ynszlyy.com